CLINICAL TRIAL: NCT01896570
Title: The Prognostic Role of Subsequent Atrial Tachycardias Occurring After Atrial Fibrillation Termination: A Prospective Randomized Trial
Brief Title: Role of Subsequent Atrial Tachycardia in Mechanisms of Persistent AF
Status: Completed | Type: Observational
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Thomas Rostock, Univ.-Prof. Dr. med., Johannes Gutenberg University Mainz
Other Study IDs: Ciritical endpoint HH
Record Dates: First submitted 2013-07-06; First posted 2013-07-11 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; catheter ablation; subsequent atrial tachycardia; mechanisms
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group A: cardioversion at AT: after achievement of AT, pts were cardioverted
- Group B: ablation to SR: After AT has been achieved, all subsequent AT were ablated with the endpoint of procedural SR termination
  Interventions: Procedure: Catheter ablation of subsequent atrial tachycardia

INTERVENTIONS:
Procedure: Catheter ablation of subsequent atrial tachycardia
  Groups: Group B: ablation to SR

SUMMARY:
In this study, the investigators aim to examine the prognostic role of subsequent Atrial Tachycardias (ATs) in the mechanisms of atrial fibrillation (AF). Therefore, the investigators compare patients who were randomly assigned to either undergo cardioversion after AF has been terminated to AT or further ablation until the achievement of sinus rhythm.

ELIGIBILITY:
Inclusion Criteria:

* persistent AF for at least 1 months,
* age > 18 years,
* refractory to drug therapy,
* no prior ablation

Exclusion Criteria:

* prior AF ablation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with persistent AF
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2009-06; Primary Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Arrhythmia-free survival | 24 months after enrolment

SECONDARY OUTCOMES:
Type of Arrhythmia recurrence | 24 months after enrolement

OTHER OUTCOMES:
Time to recurrence | after blanking period (3 months) until study end (at least 24 months)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Eppendorf, Dept. of Electrophysiology, Hamburg, Germany

REFERENCES:
- [Derived] Rostock T, Salukhe TV, Hoffmann BA, Steven D, Berner I, Mullerleile K, Theis C, Bock K, Servatius H, Sultan A, Willems S. Prognostic role of subsequent atrial tachycardias occurring during ablation of persistent atrial fibrillation: a prospective randomized trial. Circ Arrhythm Electrophysiol. 2013 Dec;6(6):1059-65. doi: 10.1161/CIRCEP.113.001019. Epub 2013 Oct 25. PMID 24162833